CLINICAL TRIAL: NCT02253576
Title: 7% Hypertonic Saline to Treat Bronchiolitis in the Emergency Department
Brief Title: Inhaled Hypertonic Saline for Bronchiolitis
Acronym: 7HSinED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not funded - never initiated
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Michael Flavin, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kuz-7HS
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Bronchiolitis
Keywords: infant; bronchiolitis; hypertonic saline
MeSH Terms: conditions — Bronchiolitis | interventions — Inhalation; Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- inhaled 7% hypertonic saline (Experimental): Three consecutive 4ml doses of 7% NaCl solution with salbutamol(0.15 mg/kg; 0.03 ml/kg of 0.5% salbutamol nebulizer solution) nebulized over a 1-hour period
  Interventions: Other: inhaled 7% hypertonic saline
- inhaled nebulized normal saline (Active Comparator): Three consecutive 4ml doses of 0.9 NaCl solution added to salbutamol(0.15 mg/kg; 0.03 ml/kg of 0.5% salbutamol nebulizer solution) nebulized over a 1-hour period
  Interventions: Other: inhaled nebulized normal saline

INTERVENTIONS:
Other: inhaled 7% hypertonic saline — Three consecutive doses of 4 ml of 7% hypertonic saline added to salbutamol, 0.15 mg/kg; 0.03 ml/kg of 0.5% salbutamol nebulizer solution over 1 hour
  Arms: inhaled 7% hypertonic saline
Other: inhaled nebulized normal saline — Three consecutive doses of 4 ml of 0.9% NaCl added to salbutamol, 0.15 mg/kg; 0.03 ml/kg of 0.5% salbutamol nebulizer solution over 1 hour
  Arms: inhaled nebulized normal saline

SUMMARY:
Study Design: This randomized, double blind, controlled, multi-centre study will occur in the Emergency Department, hospital-based Urgent Care Centre or paediatric outpatient clinics (collectively "ED") of 3 General Hospitals in Ontario and 1 in British Columbia.

DETAILED DESCRIPTION:
Children under age 2 years presenting for unscheduled care to the ED with a diagnosis of moderately severe bronchiolitis (as defined by inclusion/exclusion criteria below) will be approached for entry into the study. Recruitment will only occur when Research Assistants are on duty, is projected to include regular working hours Monday-Friday as a minimum and will continue until the calculated sample size has been obtained (anticipated 12 months). Initial routine assessment by the ED staff will identify potential subjects and Research Assistants will be notified to apply the inclusion/exclusion criteria and obtain informed consent if appropriate. Recruited subjects will be randomized to receive treatment in a double blind fashion with inhalation of nebulized study solution containing either 7% hypertonic saline (HS, study group) or 0.9% saline (NS, control group). Each dose of study solution will also contain a standard dose of bronchodilator (salbutamol, 0.15 mg/kg; 0.03 ml/kg of 0.5% salbutamol nebulizer solution) added by the ED staff. Each participant will remain on the same allocation throughout the protocol and receive 3 consecutive 4ml doses of the assigned study solution with salbutamol over a 1-hour period.

ELIGIBILITY:
Inclusion Criteria:

1. Age under 2 years
2. History of viral upper respiratory infection within previous 7 days
3. Wheezing or crackles detected on chest auscultation
4. Respiratory Distress Assessment Instrument (RDAI) score of 4 or greater or oxygen saturation (SaO2) of 94% or less in room air.

Exclusion Criteria:

History of immunodeficiency, chronic cardiopulmonary disease (other than past history of wheezing), Down syndrome, gestational age under 34 weeks.

Severe illness at presentation as defined by any of the following Respiratory rate greater than 80/min SaO2 less than 88% in room air Need for assisted ventilation Use of nebulized HS within previous 12 hours Previous enrollment in this study.

Ages: 4 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The change in respiratory distress, as measured by the Respiratory Assessment Change Score (RACS), | 120 minutes after baseline pre-treatment
  The response to treatment is determined by using the Respiratory Distress Assessment Instrument(RDAI) score and respiratory rate to calculate the Respiratory Assessment Change Score (RACS) i.e. RDAI score before minus RDAI score after treatment

SECONDARY OUTCOMES:
rates of admission to hospital | 7 days
length-of-stay of admitted patients | 28 days
rates of unscheduled return for respiratory illness to the ED | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Flavin, MD, Principal Investigator — Queen's University
Locations (3):
- Canada (3):
  - Victoria General Hospital, Victoria, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Southeastern Ontario Health Sciences Centre, Kingston, Ontario